CLINICAL TRIAL: NCT00351780
Title: Physiologic Evaluation of the Provisional Side Branch Intervention Strategy for Bifurcation Lesions Using Fractional Flow Reserve
Brief Title: Fractional Flow Reserve-guided Provisional Side Branch Intervention
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Seoul National University Hospital, Seoul National University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-0602-027-167
Record Dates: First submitted 2006-07-12; First posted 2006-07-13 (Estimated); Last update posted 2011-07-18 (Estimated); Status verified 2011-07

CONDITIONS: Coronary Artery Disease
Keywords: fractional flow reserve; bifurcation; stent
MeSH Terms: conditions — Coronary Artery Disease

INTERVENTIONS:
Device: FFR measurement, side branch angioplasty

SUMMARY:
Study purpose: To evaluate fractional flow reserve-guided side branch intervention strategy Method: Provisional side branch intervention if jailed side branch FFR<0.75

DETAILED DESCRIPTION:
Patients with de novo, coronary bifurcation lesions with jailed side branches after successful drug-eluting stent implantation at the main branches will be prospectively and consecutively enrolled. Control group patients will be selected from the database.

Jailed side branches need to have an ostial stenosis >50%, vessel size >2 mm, vessel length >40 mm and lesion length <10 mm by visual estimation.

Study procedure Coronary stenting of the main branch should be performed with standard interventional techniques using drug-eluting stents. In the FFR group, pressure measurement would be performed using a 0.014 inch pressure guide wire (PressureWire, Radi Medical Systems, Uppsala, Sweden)Lesions with an FFR <0.75 are considered to have functionally significant stenosis and side branch balloon dilatation is allowed only for these lesions. It is recommended to use a smaller balloon than the side branch vessel diameter. After kissing balloon inflation, FFR will be measured again at the same site and further intervention is only recommended when FFR was <0.75 after kissing balloon dilatation. In the conventional group, the decision to treat the side branch lesion and the method of intervention are all up to the operators' discretion.

ELIGIBILITY:
Inclusion Criteria:

Jailed side branches with an ostial stenosis >50%, vessel size >2mm, vessel length >40mm and lesion length <10mm by visual estimation.

Exclusion Criteria:

ST elevation myocardial infarction Left main stenosis, totally occluded lesion Angiographically visible thrombus, significant lesion within the main branch proximal to the stented segment, significant distal lesion at a side branch Regional wall motion abnormalities of the stented artery and jailed side branch segments Left ventricular ejection fraction<40% Primary myocardial disease Serum creatinine >2mg/dl Predilatation of side branch before the main branch stent implantation Contraindications to adenosine

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2004-06; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bon-Kwon Koo, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea